CLINICAL TRIAL: NCT03896750
Title: A Phase 1, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics and Safety of Pretomanid in Participants With Renal Impairment Compared to Participants With Normal Renal Function
Brief Title: Single-Dose Study to Evaluate the PKs of Pretomanid in Participants With Renal Impairment Compared to Participants With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-0037
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-07-08

CONDITIONS: Renal Impairment; Tuberculosis
Keywords: Open-Label; Pretomanid; Renal Pharmacokinetic; Single-Dose
MeSH Terms: conditions — Renal Insufficiency; Tuberculosis | interventions — pretomanid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part A Group 1A (Active Comparator): 6 healthy participants with normal renal function: Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR > / = 90 mL/min) matched to Group 2 by race, gender, age (+/- 10 years, but between 18 to 85 years of age) and body mass index (BMI) (18 to 40 kg/m^2) will receive a single oral dose of 200 mg pretomanid
  Interventions: Drug: PA-824
- Part A Group 2 (Experimental): 6 participants with severe renal impairment: Stage 4, Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR 15-29 mL/min), and End Stage Renal Disease (ESRD) not on dialysis: Stage 5, Modification of Diet in Renal Disease (MDRD) with estimated Glomerular Filtration Rate (eGFR < 15 mL/min) matched to Group 1A will receive a single oral dose of 200 mg pretomanid
  Interventions: Drug: PA-824
- Part B Group 1B (Active Comparator): 6 healthy participants with Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR of > / = 90 mL/min) matched to Group 3 by race, gender, age (+/- 10 years, but between 18 to 85 years of age) and body mass index (BMI) (18 to 40 kg/m^2) will receive a single oral dose of 200 mg pretomanid after the PK and safety of subjects enrolled in Part A have been reviewed
  Interventions: Drug: PA-824
- Part B Group 1C (Active Comparator): 6 healthy participants: with Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR > / = 90 mL/min) matched to Group 4 by race, gender, age (+/- 10 years, but between 18 to 85 years of age) and body mass index (BMI) (18 to 40 kg/m^2) will receive a single oral dose of 200 mg pretomanid after the PK and safety of subjects enrolled in Part A have been reviewed
  Interventions: Drug: PA-824
- Part B Group 3 (Experimental): 6 participants with mild renal impairment: Stage 2, Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR 60-89 mL/min) matched to Group 1B will receive a single oral dose of 200 mg pretomanid after the PK and safety of subjects enrolled in Part A have been reviewed
  Interventions: Drug: PA-824
- Part B Group 4 (Experimental): 6 participants with moderate renal impairment: Stage 3, Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR = 30-59 mL/min) matched to Group 1C will receive a single oral dose of 200 mg pretomanid after the PK and safety of subjects enrolled in Part A have been reviewed
  Interventions: Drug: PA-824

INTERVENTIONS:
Drug: PA-824 — PA-824, a nitroimidazooxazine, used in prior studies of pretomanid is a novel TB treatment that is being investigated for use with other TB drugs to shorten and/or simplify regimens to treat either drug susceptible or resistant disease. After fasting for a minimum of 8 hours, subjects will receive one dose of 200 mg of pretomanid orally under direct supervision with 240 mL of water and a mouth check will be done.

SUMMARY:
This is a Phase 1, open-label, single-dose, sequential group study to compare the safety and pharmacokinetics (PK) of pretomanid in the following groups of participants: 1) participants with severe renal impairment including those with end stage renal disease (ESRD) not on dialysis, and participants with mild or moderate renal impairment, designated as Groups 2, 3, and 4, respectively; and 2) participants with normal renal function matched to the above renal impairment groups, designated as Groups 1A, 1B, and 1C, respectively.

The study will be conducted following a reduced PK study design in Part A. Part A will enroll participants from Group 1A (i.e., 6 healthy matched controls) and Group 2 (i.e., 6 participants with severe renal impairment and ESRD, not on dialysis). A decision to proceed to Part B will be made after the PK of pretomanid, and safety in participants enrolled in Part A have been reviewed. If Part A demonstrates at least a 50% increase in pretomanid area under the plasma concentration-time curve (AUC) in Group 2 (severe renal impairments and ESRD, not on dialysis) relative to the exposures in Group 1A (matched participants with normal renal function), then the reduced PK study will extend to the full PK study to enroll participants into Part B (i.e., to investigate mild and moderate renal impairment). All Part B groups (1B, 1C, 3, and 4) will be enrolled concurrently.

If the reduced PK study shows at least a 50% increase in AUC in patients with severe renal impairment and patients with ESRD not yet on dialysis relative to the matched healthy controls, a "full PK" renal impairment study in patients with all intermediate levels of renal function impairment should be conducted. Otherwise, no further study is recommended.

The approximate patient involvement will be 3 months. The primary objective is to evaluate the PK profiles of pretomanid in plasma and urine after a single oral dose of 200 mg in participants with renal impairment compared to matched healthy controls.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-dose, sequential group study to compare the safety and pharmacokinetics (PK) of pretomanid in the following groups of participants: 1) participants with severe renal impairment including those with end stage renal disease (ESRD) not on dialysis, and participants with mild or moderate renal impairment, designated as Groups 2, 3, and 4, respectively; and 2) participants with normal renal function matched to the above renal impairment groups, designated as Groups 1A, 1B, and 1C, respectively.

The study will be conducted following a reduced PK study design in Part A. Part A will enroll participants from Group 1A (i.e., 6 healthy matched controls) and Group 2 (i.e., 6 participants with severe renal impairment and ESRD, not on dialysis). A decision to proceed to Part B will be made after the PK of pretomanid, and safety in participants enrolled in Part A have been reviewed. If Part A demonstrates at least a 50% increase in pretomanid area under the plasma concentration-time curve (AUC) in Group 2 (severe renal impairments and ESRD, not on dialysis) relative to the exposures in Group 1A (matched participants with normal renal function), then the reduced PK study will extend to the full PK study to enroll participants into Part B (i.e., to investigate mild and moderate renal impairment). All Part B groups (1B, 1C, 3, and 4) will be enrolled concurrently.

If the reduced PK study shows at least a 50% increase in AUC in patients with severe renal impairment and patients with ESRD not yet on dialysis relative to the matched healthy controls, a "full PK" renal impairment study in patients with all intermediate levels of renal function impairment should be conducted. Otherwise, no further study is recommended.

The approximate patient involvement will be 3 months. The primary objective is to evaluate the PK profiles of pretomanid in plasma and urine after a single oral dose of 200 mg in participants with renal impairment compared to matched healthy controls. The secondary objectives are 1) to assess the safety profile of a single oral dose of 200 mg pretomanid in renally impaired participants to matched healthy controls; and 2) to evaluate the PK profiles or representative pretomanid metabolites (M19 and M50) in plasma and urine.

ELIGIBILITY:
Inclusion Criteria:

Participant Inclusion Criteria for Patients with Renal Impairment (Groups 2-4)

1. Have the ability to understand the requirements of the study and have provided written informed consent* before any study-related procedure is performed.

   *As evidence by signature on an informed consent document approved by the Institutional Review Board
2. Agree to abide by the study restrictions.
3. Are between the ages of 18 and 85 years, inclusive, at the time of enrollment.
4. Must have mild, moderate, or severe renal impairment or end stage renal disease (ESRD), but are not on dialysis.
5. Have no history of chronic tobacco/nicotine usage (i.e., >10 cigarettes per day for 3 months minimum prior to admission).
6. Have corrected QT interval by Fridericia (QTcF) <460 msec on Electrocardiogram (ECG).
7. Have a Body Mass Index (BMI) of 18 to 40 kg/m^2 at enrollment.
8. Women of childbearing potential** must use an acceptable contraception method*** for the duration of the study.

   **Not sterilized via tubal ligation, bilateral oophorectomy, bilateral salpingectomy, hysterectomy, implanted contraceptive device placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses if menopausal.

   ***Includes, non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the participant receiving study product, barrier methods such as condoms with spermicide or diaphragms/cervical caps with spermicide, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").
9. If participant is male and capable of reproduction, agrees to avoid fathering a child for the duration of the study by using an acceptable method of birth control****.

   ****In addition to the use of a barrier method (condom) unless vasectomized, acceptable methods of birth control are restricted to a monogamous relationship with a woman who agrees to use acceptable contraception as outlined in inclusion criterion #8, and/or abstinence from sexual intercourse with women.
10. Women of childbearing potential must have a negative urine pregnancy test within 24 hours prior to receipt of study product.

Participant Inclusion Criteria for Healthy Participants (Groups 1A-1C)

1. Have the ability to understand the requirements of the study and have provided written informed consent* before any study-related procedure is performed.

   *As evidence by signature on an informed consent document approved by the Institutional Review Board (IRB).
2. Agree to abide by the study restrictions.
3. Are healthy male or non-pregnant female, between the ages of 18 and 85 years, inclusive, with normal GFR >90 at screening.
4. Have no history of chronic tobacco/nicotine usage (i.e., >10 cigarettes per day for 3 months minimum prior to admission).
5. Have a normal corrected QT interval by Fridericia (QTcF) <460 msec on ECG.
6. Have a Body Mass Index of 18 to 40 kg/m^2 at enrollment.
7. Women of childbearing potential** must use an acceptable contraception method*** for the duration of the study.

   **Not sterilized via tubal ligation, bilateral oophorectomy, bilateral salpingectomy, hysterectomy, implanted contraceptive device placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses if menopausal.

   ***Includes non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the participant receiving study product, barrier methods such as condoms with spermicide or diaphragms/cervical caps with spermicide, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").
8. If participant is male and capable of reproduction, agrees to avoid fathering a child for the duration of the study by using an acceptable method of birth control****.

   ****In addition to the use of a barrier method (condom) unless vasectomized, acceptable methods of birth control are restricted to a monogamous relationship with a woman who agrees to use acceptable contraception as outlined in inclusion criterion #7, and/or abstinence from sexual intercourse with women.
9. Women of childbearing potential must have a negative urine pregnancy test within 24 hours prior to receipt of study product.

Exclusion Criteria:

Participant Exclusion Criteria for Patients with Renal Impairment (Groups 2-4)

1. History of known active TB.
2. History of peptic ulcer disease.
3. Known hypersensitivity to pretomanid or any of the excipients.
4. History of any clinically significant uncontrolled cardiac abnormality (as deemed by the Principal Investigator (PI)).
5. Any clinically significant electrocardiogram (ECG) abnormality at screening*.

   *Note: the following can be considered not clinically significant:

   - Heart rate </= 50 beats per minute (bpm) (sinus bradycardia with heart rate between 45 and 49, inclusive, is acceptable only in younger athletic participants, as determined by the Principal Investigator ))
   * Mild first-degree atrioventricular (A-V) block (P-R interval >0.23 seconds)
   * Right or left axis deviation
   * Incomplete right bundle branch block
   * Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic participants
6. History of, or screening results show a corrected QT interval by Fridericia (QTcF) >/= 460 msec.
7. Family history of Long-QT Syndrome or sudden death when a cause of death is unknown.
8. Inability to swallow tablets.
9. History of fever or documented fever (oral temperature >/= 100.4 degrees F) in the 48 hours prior to admission to the hospital.
10. Resting pulse rate <50 or >110 bpm at Screening.
11. At Screening, blood pressure >/= 20 mm Hg systolic or >10 mm Hg diastolic above baseline** (sitting).

    **Baseline is most recent blood pressure in the last 3 months.
12. Current hyperkalemia or hypomagnesemia.
13. Positive result of urine drug screen or blood alcohol screen prior to hospital admission except for approved prescriptions that are not opiates and benzodiazepines.
14. Significant history of drug and/or food allergies (as deemed by the Principal Investigator (PI)).
15. For women, participant is pregnant (positive test for urine Human Chorionic Gonadotropin [HCG]) at screening or Admission, breastfeeding, or planning to conceive for the duration of the study.
16. Any contraindication to the use of nitroimidazoles, or prior treatment with pretomanid or delamanid.
17. Treatment with strong or moderate CYP3A4 inducers or inhibitors*** within 14 days before admission and during the study****.

    ***Except hormonal contraceptives

    ****In the opinion of the site investigator
18. Use of St. John's Wort within 7 days prior to admission and during the entire study.
19. Consumption of products containing grapefruit within 5 days prior to dosing until Visit 01N.
20. Donation of whole blood or blood products >500 mL within 30 days from screening and/or plans to donate during the study or up to 14 days after dosing.
21. Participation in another interventional clinical trial within 30 days prior to dosing until after the last study visit.
22. Hemoglobin (Hgb) <8.0 g/dL in both men and women at the screening visit.
23. Positive Screening test for Hepatitis C Virus (HCV), Hepatitis B Virus (HBV), or Human Immunodeficiency Virus (HIV).
24. Renal transplant.
25. Scheduled for hemodialysis or peritoneal dialysis.
26. Presence of any condition or finding***** which would jeopardize participant safety, impact study result validity, or diminish the participant's ability to undergo all study procedures and assessments.

    *****In the opinion of the investigator
27. For men, semen donation for the duration of the study.
28. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) > 2.5 x Upper Limit of Normal (ULN).
29. Hyperbilirubinemia >1.5 x Upper Limits of Normal (ULN).

Participant Exclusion Criteria for Healthy Participants (Groups 1A-1C)

1. History of known active TB.
2. History of peptic ulcer disease.
3. Known hypersensitivity to pretomanid or any of the excipients.
4. History of any clinically significant uncontrolled cardiac abnormality (as deemed by the Principal Investigator (PI)).
5. Any clinically significant ECG abnormality at screening.*

   *Note: the following can be considered not clinically significant:
   * Heart rate </= 50 bpm (sinus bradycardia with heart rate between 45 and 49, inclusive, is acceptable only in younger athletic participants)
   * Mild first-degree A-V block (P-R interval >0.23 seconds)
   * Right or left axis deviation
   * Incomplete right bundle branch block
   * Isolated left anterior fascicular block (left anterior hemiblock) in younger athletic participants
6. Family history of Long-QT Syndrome or sudden death when a cause of death is unknown.
7. Inability to swallow tablets.
8. History of fever or documented fever (oral temperature >/= 100.4 degrees F) in the 48 hours prior to admission to the hospital.
9. At Screening blood pressure >140/90 mm Hg or <90/65 mm Hg (sitting).
10. History of, or screening results show a corrected QT interval by Fridericia (QTcF) >460 msec.
11. Positive result of urine drug screen or blood alcohol screen prior to hospital admission except for approved prescriptions that are not opiates and benzodiazepines.
12. Significant history of drug and/or food allergies (as deemed by the Principal Investigator (PI)).
13. Women of childbearing potential with a positive urine pregnancy test within 24 hours prior to receipt of study product.
14. Any contraindication to the use of nitroimidazoles, or prior treatment with pretomanid or delamanid.
15. Treatment with strong or moderate CYP3A4 inducers or inhibitors** within 14 days before admission and during the study***.

    **Except hormonal contraceptives

    ***In the opinion of the site Principal Investigator (PI)
16. Use of St. John's Wort within 7 days prior to admission and during the entire study.
17. Consumption of products containing grapefruit within 5 days prior to dosing until Visit 01N.
18. Donation of whole blood or blood products >500 mL within 30 days from screening and/or plans to donate during the study or up to 14 days after dosing.
19. Participation in another interventional clinical trial within 30 days prior to dosing until after the last study visit.
20. Hgb <10.0 g/dL in both men and women at the screening visit.
21. Positive Screening test for Hepatitis C virus (HCV), Hepatitis B virus (HBV), or Human Immunodeficiency Virus (HIV).
22. Renal transplant.
23. Presence of any condition or finding**** which would jeopardize participant safety, impact study result validity, or diminish the participant's ability to undergo all study procedures and assessments.

    ****In the opinion of the investigator
24. For men, semen donation for the duration of the study.
25. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) > Upper Limits of Normal (ULN).
26. Bilirubin > Upper Limits of Normal (ULN)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Advanced Pharma - Miami, Miami, Florida
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - Alliance for Multispecialty Research, LLC - Knoxville, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population was represented by participants of varying degrees of renal disease, recruited from the community at large. Participants were between 18 and 85 years, inclusive at the time of enrollment. Enrollment occurred from 17APR2024 to 05AUG2024.
Groups:
- Part A Group 1A - Healthy Matched Controls: Healthy participants with normal renal function: Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR > / = 90 mL/min) matched to Group 2 by race, gender, age (+/- 10 years, but between 18 to 85 years of age) and body mass index (BMI) (18 to 40 kg/m^2) will receive a single oral dose of 200 mg pretomanid
  PA-824: PA-824, a nitroimidazooxazine, used in prior studies of pretomanid is a novel TB treatment that is being investigated for use with other TB drugs to shorten and/or simplify regimens to treat either drug susceptible or resistant disease. After fasting for a minimum of 8 hours, subjects will receive one dose of 200 mg of pretomanid orally under direct supervision with 240 mL of water and a mouth check will be done.
- Part A Group 2 - ESRD Not on Dialysis: Participants with End Stage Renal Disease (ESRD) not on dialysis: Stage 5, Modification of Diet in Renal Disease (MDRD) with estimated Glomerular Filtration Rate (eGFR < 15 mL/min) matched to Group 1A will receive a single oral dose of 200 mg pretomanid
  PA-824: PA-824, a nitroimidazooxazine, used in prior studies of pretomanid is a novel TB treatment that is being investigated for use with other TB drugs to shorten and/or simplify regimens to treat either drug susceptible or resistant disease. After fasting for a minimum of 8 hours, subjects will receive one dose of 200 mg of pretomanid orally under direct supervision with 240 mL of water and a mouth check will be done.
- Part A Group 2 - Severe Renal Impairment: Participants with severe renal impairment: Stage 4, Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR 15-29 mL/min) matched to Group 1A will receive a single oral dose of 200 mg pretomanid
  PA-824: PA-824, a nitroimidazooxazine, used in prior studies of pretomanid is a novel TB treatment that is being investigated for use with other TB drugs to shorten and/or simplify regimens to treat either drug susceptible or resistant disease. After fasting for a minimum of 8 hours, subjects will receive one dose of 200 mg of pretomanid orally under direct supervision with 240 mL of water and a mouth check will be done.
- Part B Group 3 - Mild Renal Impairment: Participants with mild renal impairment: Stage 2, Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR 60-89 mL/min) matched to Group 1B will receive a single oral dose of 200 mg pretomanid after the PK and safety of subjects enrolled in Part A have been reviewed
  PA-824: PA-824, a nitroimidazooxazine, used in prior studies of pretomanid is a novel TB treatment that is being investigated for use with other TB drugs to shorten and/or simplify regimens to treat either drug susceptible or resistant disease. After fasting for a minimum of 8 hours, subjects will receive one dose of 200 mg of pretomanid orally under direct supervision with 240 mL of water and a mouth check will be done.
- Part B Group 4 - Moderate Renal Impairment: Participants with moderate renal impairment: Stage 3, Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR = 30-59 mL/min) matched to Group 1C will receive a single oral dose of 200 mg pretomanid after the PK and safety of subjects enrolled in Part A have been reviewed
  PA-824: PA-824, a nitroimidazooxazine, used in prior studies of pretomanid is a novel TB treatment that is being investigated for use with other TB drugs to shorten and/or simplify regimens to treat either drug susceptible or resistant disease. After fasting for a minimum of 8 hours, subjects will receive one dose of 200 mg of pretomanid orally under direct supervision with 240 mL of water and a mouth check will be done.
Period: Overall Study
Arm/Group | Part A Group 1A - Healthy Matched Controls | Part A Group 2 - ESRD Not on Dialysis | Part A Group 2 - Severe Renal Impairment | Part B Group 3 - Mild Renal Impairment | Part B Group 4 - Moderate Renal Impairment
Started | 6 | 1 | 5 | 0 | 0
Completed | 6 | 1 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Matched Controls: Healthy participants with normal renal function received a single oral dose of 200 mg pretomanid
- ESRD Not on Dialysis: Participants with End Stage Renal Disease (ESRD) not on dialysis received a single oral dose of 200 mg pretomanid
- Severe Renal Impairment: Participants with severe renal impairment received a single oral dose of 200 mg pretomanid
- Total: Total of all reporting groups
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment | Total
Number analyzed (Participants) | 6 | 1 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (12.8) | 40.0 | 62.0 (10.0) | 56.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 6
  Male | 3 | 0 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 1 | 7
  Not Hispanic or Latino | 1 | 0 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 5 | 1 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 1 | 5 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.17 (2.84) | 40.0 | 36.02 (3.42) | 34.43 (3.83)
Height [Mean (Standard Deviation); unit: cm] | 163.55 (8.85) | 155.00 | 167.42 (3.61) | 164.45 (7.27)
Weight [Mean (Standard Deviation); unit: kg] | 86.62 (15.15) | 96.00 | 101.12 (11.53) | 93.44 (14.34)

OUTCOME MEASURES:

1. Primary Outcome: Fold Change in Pretomanid AUC(0-last) in Participants With Renal Impairment as Compared to Matched Healthy Controls
Description: The mean fold change of AUC(0-last) Area under the concentration time-curve to the last concentration above the lower limit of quantitation at specified pre-dose and post-dose time points was calculated by noncompartmental analysis using the linear up log down method. The mean fold change of each enrolled renal impairment arm as compared to the Healthy Matched Control arm was calculated by a linear regression model controlling for site.
Time Frame: Day 1 at 1, 2, 4, 5, 6, 8, 12, 16 hours post dose; Day 2 at 24 and 36 hours post dose; Day 3 at 48 hours post dose; Day 4 at 72 hours post dose; and Day 5 at 96 hours post dose.
Population: The PK plasma analysis subset consisted of all participants with sufficient plasma PK data available to estimate the plasma PK parameters using noncompartmental methods.
Measure: Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
ng*h/mL | 77130 [62810 to 91460] | 63600 | 62660 [54280 to 71040]
Statistical Analysis 1: Comparison: ESRD Not on Dialysis; No formal hypothesis testing was conducted. Assuming a 20% coefficient of variation for the AUC(0-last) of both groups, the probability of observing at least a 50% increase in the geometric mean ratio of AUCs given a true 100% increase is >99%. The probability of the lower bound of the 90% CI for the geometric mean ratio of AUCs being at least 1.5 in this scenario is approximately 70%; Test type: Equivalence — Equivalence analysis by 90% confidence interval. If the interval encompasses 1 there is no clinically meaningful difference in pretomanid AUC(0-last). Assuming a 20% coefficient of variation for the AUC(0-last) of both groups, the probability of observing at least a 50% increase in the geometric mean ratio of AUCs given a true 100% increase is >99%. The probability of the lower bound of the 90% CI for the geometric mean ratio of AUCs being at least 1.5 in this scenario is approximately 70%; Regression, Linear; Adjusted for site; Mean Ratio = 0.83, 90% CI 2-sided [0.54 to 1.26]
Statistical Analysis 2: Comparison: Severe Renal Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Regression, Linear; Adjusted for site; Mean Ratio = 0.87, 90% CI 2-sided [0.67 to 1.14]

2. Primary Outcome: Fold Change in Pretomanid AUC(0-infinity) in Participants With Renal Impairment as Compared to Matched Healthy Controls
Description: The mean fold change of AUC(0-infinity) was calculated by noncompartmental analysis using the linear up log down method with the area extrapolated to infinity as Clast/Lambda_z where Clast was the last observed concentration and Lambda_z is the elimination rate constant. The mean fold change of each enrolled renal impairment arm as compared to the Healthy Matched Control arm was calculated by a linear regression model controlling for site.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: ng*h/mL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
ng*h/mL | 88650 [69340 to 108000] | 76400 | 76740 [66610 to 86870]
Statistical Analysis 1: Comparison: ESRD Not on Dialysis; No formal hypothesis testing was conducted. Assuming a 20% coefficient of variation for the AUC(0-infinity) of both groups, the probability of observing at least a 50% increase in the geometric mean ratio of AUCs given a true 100% increase is >99%. The probability of the lower bound of the 90% CI for the geometric mean ratio of AUCs being at least 1.5 in this scenario is approximately 70%; Test type: Equivalence — Equivalence analysis by 90% confidence interval. If the interval encompasses 1 there is no clinically meaningful difference in pretomanid AUC(0-infinity). Assuming a 20% coefficient of variation for the AUC(0-infinity) of both groups, the probability of observing at least 50% increase in the geometric mean ratio of AUCs given a true 100% increase is >99%. The probability of the lower bound of the 90% CI for the geometric mean ratio of AUCs being at least 1.5 in this scenario is approximately 70%; Regression, Linear; Adjusted for site; Mean Ratio = 0.87, 90% CI 2-sided [0.54 to 1.39]
Statistical Analysis 2: Comparison: Severe Renal Impairment; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Regression, Linear; Adjusted for site; Mean Ratio = 0.95, 90% CI 2-sided [0.71 to 1.28]

3. Secondary Outcome: Area Under the M19 and M50 Concentration Time-curve Extrapolated to Infinity at Specified Pre-dose and Post-dose Time Points
Description: AUC(0-infinity) was calculated by noncompartmental analysis using the linear up log down method with the area extrapolated to infinity as Clast/Lambda_z where Clast was the last observed concentration and Lambda_z is the elimination rate constant. M19 and M50 are the two primary representative metabolites of pretomanid.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
ng*h/mL
  M19 | 4013 (2021) | 5980 | 7458 (4410)
  M50 | 700.7 (251.3) | 737.0 | 1132 (547.1)

4. Secondary Outcome: Area Under the M19 and M50 Concentration Time-curve to the Last Concentration Above the Lower Limit of Quantitation at Specified Pre-dose and Post-dose Time Points
Description: AUC(0-last) Area under the concentration time-curve to the last concentration above the lower limit of quantitation at specified pre-dose and post-dose time points was calculated by noncompartmental analysis using the linear up log down method. M19 and M50 are the two primary representative metabolites of pretomanid.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
ng*h/mL
  M19 | 3503 (1852) | 4150 | 4746 (3064)
  M50 | 585.0 (202.5) | 631.0 | 932.8 (479.7)

5. Secondary Outcome: Maximum M19 and M50 Concentrations at Specified Pre-dose and Post-dose Time Points
Description: Maximum M19 and M50 concentrations is the maximum observed drug concentration in blood plasma at specified pre-dose and post-dose timepoints. M19 and M50 are the two primary representative metabolites of pretomanid.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
ng/mL
  M19 | 82.05 (33.34) | 81.30 | 73.66 (48.38)
  M50 | 15.05 (3.603) | 12.60 | 16.28 (8.149)

6. Secondary Outcome: Apparent Terminal Elimination Half-life of M19 and M50 at Specified Pre-dose and Post-dose Time Points
Description: Apparent terminal half-life of M19 and M50 at specified pre-dose and post-dose timepoints was estimated by ln(2)/Lambda_z, where Lambda_z is the elimination rate constant. M19 and M50 are the two primary representative metabolites of pretomanid.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
Hours
  M19 | 31.58 (8.06) | 48.80 | 53.68 (14.29)
  M50 | 31.12 (7.13) | 31.0 | 35.68 (5.97)

7. Secondary Outcome: Renal Clearance of M19 and M50 at Specified Pre-dose and Post-dose Time Points
Description: Renal clearance (CLr) of M19 and M50 calculated as the amount excreted in urine to time t in urine divided by the plasma AUC from 0 to time t. M19 and M50 are the two primary representative metabolites of pretomanid.
Time Frame: as for outcome 1
Population: The PK urine analysis subset will consist of all participants with sufficient urine PK data available to estimate the urine PK parameters.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
L/h
  M19 | 0.222 (0.134) | 0.170 | 0.440 (0.567)
  M50 | 5.935 (3.857) | 0.930 | 0.634 (0.139)

8. Secondary Outcome: Amount of M19 and M50 Excreted in Urine at Specified Pre-dose and Post-dose Time Points
Description: Amount of M19 and M50 excreted in Urine [Ae(0-t)] is the sum of the amount of M19 and M50 recovered in urine during the collection window. M19 and M50 are the two primary representative metabolites of pretomanid.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ug
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
ug
  M19 | 678.3 (314.0) | 715.0 | 1637 (1894)
  M50 | 3302 (2420) | 585.0 | 548.0 (143.4)

9. Secondary Outcome: Apparent Volume of Distribution of M19 and M50 at Specified Pre-dose and Post-dose Time Points
Description: Apparent Volume of Distribution at specified pre-dose and post-dose timepoints is the volume that the total amount of administered drug would occupy to provide the same concentration as it currently is in blood plasma divided by the bioavailability. It is calculated by Dose/[Lambda_z x AUC(0-infinity)]. M19 and M50 are the two primary representative metabolites of pretomanid.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
L
  M19 | 2793 (1414) | 2350 | 3106 (2543)
  M50 | 13570 (3050) | 12100 | 10540 (4333)

10. Secondary Outcome: Time of Maximum M19 and M50 Concentration at Specified Pre-dose and Post-dose Time Points
Description: Time of maximum M19 and M50 concentration (Tmax) at specified pre-dose and post-dose timepoints. M19 and M50 are the two primary representative metabolites of pretomanid.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
Hours
  M19 | 10.67 (7.45) | 24.00 | 22.42 (15.43)
  M50 | 7.50 (3.78) | 16.00 | 13.60 (2.19)

11. Secondary Outcome: Apparent Oral Clearance of M19 and M50 From Dose/AUC(0-infinity) at Specified Pre-dose and Post-dose Time Points
Description: Apparent oral clearance was calculated by noncompartmental analysis using the formula Dose/AUC(0-infinity). M19 and M50 are the two primary representative metabolites of pretomanid.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
L/h
  M19 | 59.73 (24.27) | 33.40 | 36.50 (24.10)
  M50 | 318.8 (116.5) | 272.0 | 200.5 (62.07)

12. Secondary Outcome: Number of Participants With and Severity of Adverse Events
Description: An Adverse Event (AE) was defined as any unfavorable or unintended medical occurrence temporally associated with the use of a study drug, device, other medical product, or procedure whether or not it is considered related to the product itself.
Time Frame: Day 1 to Day 85
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
Participants
  Lab finding of Mild or Worse Severity Through Day 12 | 0 | 1 | 5
  Unsolicited AEs | 0 | 0 | 3
  Unsolicited Treatment Emergent AEs | 0 | 0 | 3
  Mild Related Unsolicited Treatment Emergent AEs | 0 | 0 | 2
  Moderate Related Unsolicited Treatment Emergent AEs | 0 | 0 | 1

13. Secondary Outcome: Mean Change From Baseline in Alanine Aminotransferase (ALT)
Description: The mean change from baseline was calculated by taking the mean of each participant value at the specified day minus the value last recorded prior to drug administration.
Time Frame: Day 5 and Day 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
U/L
  Day 5 | 0.0 (5.5) | 2.0 | 2.0 (8.2)
  Day 12 | 1.2 (6.1) | 1.0 | 4.0 (7.6)

14. Secondary Outcome: Mean Change From Baseline in Aspartate Aminotransferase (AST)
Description: as for outcome 13
Time Frame: Day 5 and Day 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
U/L
  Day 5 | -2.3 (4.6) | 1.0 | 0.4 (1.5)
  Day 12 | 0.5 (3.3) | -2.0 | 0.8 (2.5)

15. Secondary Outcome: Mean Change From Baseline in Blood Urea Nitrogen (BUN)
Description: as for outcome 13
Time Frame: Day 5 and Day 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
mg/dL
  Day 5 | -1.5 (4.5) | 2.0 | 6.6 (19.6)
  Day 12 | -1.2 (2.5) | -9.0 | 3.0 (23.0)

16. Secondary Outcome: Mean Change From Baseline in Creatinine
Description: as for outcome 13
Time Frame: Day 5 and Day 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
mg/dL
  Day 5 | 0.032 (0.097) | -0.520 | 0.330 (0.738)
  Day 12 | -0.017 (0.108) | -0.400 | 0.028 (0.448)

17. Secondary Outcome: Mean Change From Baseline in Hemoglobin (Hgb)
Description: as for outcome 13
Time Frame: Day 5 and Day 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
g/dL
  Day 5 | 0.52 (0.83) | -0.60 | -0.66 (0.85)
  Day 12 | -0.37 (0.67) | 0.00 | -1.26 (0.65)

18. Secondary Outcome: Mean Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: as for outcome 13
Time Frame: Day 5 and Day 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
mL/min/1.73m^2
  Day 5 | -6.0 (19.9) | 4.0 | -2.6 (5.5)
  Day 12 | 3.2 (20.4) | 1.0 | 0.6 (2.6)

19. Secondary Outcome: Mean Change From Baseline in Magnesium
Description: as for outcome 13
Time Frame: Day 5 and Day 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
mg/dL
  Day 5 | -0.12 (0.20) | -0.20 | -0.10 (0.22)
  Day 12 | 0.00 (0.14) | -0.20 | -0.04 (0.23)

20. Secondary Outcome: Mean Change From Baseline in Serum Potassium
Description: as for outcome 13
Time Frame: Day 5 and Day 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
mmol/L
  Day 5 | 0.27 (0.46) | 0.60 | 0.18 (0.42)
  Day 12 | 0.12 (0.29) | 0.10 | 0.14 (0.71)

21. Secondary Outcome: Mean Change From Baseline in Total Bilirubin
Description: as for outcome 13
Time Frame: Day 5 and Day 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
mg/dL
  Day 5 | 0.03 (0.27) | 0.00 | -0.02 (0.25)
  Day 12 | 0.10 (0.31) | 0.00 | -0.02 (0.15)

22. Secondary Outcome: Mean Change in Oral Temperature From Baseline
Description: as for outcome 13
Time Frame: Days 1, 2, 3, 4, 5, and 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
degrees Fahrenheit
  Day 1 (12 hours post-dose) | -0.07 (0.31) | -0.90 | 0.14 (0.54)
  Day 2 (24 hours post-dose) | -0.12 (0.15) | -0.50 | -0.22 (0.24)
  Day 3 (48 hours post-dose) | -0.10 (0.26) | -0.20 | 0.20 (0.53)
  Day 4 (72 hours post-dose) | -0.22 (0.31) | -0.20 | -0.24 (0.34)
  Day 5 (96 hours post-dose) | -0.28 (0.42) | -0.70 | -0.06 (0.21)
  Day 12 | -0.22 (0.29) | -1.20 | 0.02 (0.16)

23. Secondary Outcome: Mean Change in Pulse From Baseline
Description: as for outcome 13
Time Frame: Days 1, 2, 3, 4, 5, and 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
bpm
  Day 1 (12 hours post-dose) | -0.3 (8.3) | -8.0 | 0.4 (5.0)
  Day 2 (24 hours post-dose) | 3.7 (6.7) | -3.0 | -0.2 (5.2)
  Day 3 (48 hours post-dose) | 3.5 (3.3) | -6.0 | -1.4 (6.5)
  Day 4 (72 hours post-dose) | 5.7 (7.9) | -18.0 | -4.2 (3.8)
  Day 5 (96 hours post-dose) | 2.0 (7.6) | -18.0 | -1.8 (4.8)
  Day 12 | 5.3 (5.6) | -4.0 | -6.8 (6.1)

24. Secondary Outcome: Mean Change in Sitting Systolic Blood Pressure From Baseline
Description: as for outcome 13
Time Frame: Days 1, 2, 3, 4, 5, and 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
mmHg
  Day 1 (12 hours post-dose) | 0.8 (4.4) | -4.0 | 2.0 (19.2)
  Day 2 (24 hours post-dose) | -6.5 (7.5) | -16.0 | -15.0 (14.9)
  Day 3 (48 hours post-dose) | 0.3 (10.1) | -23.0 | -11.2 (14.0)
  Day 4 (72 hours post-dose) | 0.8 (8.1) | -20.0 | -3.4 (17.7)
  Day 5 (96 hours post-dose) | 0.5 (6.9) | -17.0 | -3.8 (13.5)
  Day 12 | 0.8 (4.8) | -13.0 | -5.4 (20.2)

25. Secondary Outcome: Mean Change in Sitting Diastolic Blood Pressure From Baseline
Description: as for outcome 13
Time Frame: Days 1, 2, 3, 4, 5, and 12
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
mmHg
  Day 1 (12 hours post-dose) | 1.3 (2.5) | 3.0 | 2.0 (9.8)
  Day 2 (24 hours post-dose) | -3.7 (6.3) | -6.0 | -2.4 (7.0)
  Day 3 (48 hours post-dose) | -0.5 (6.7) | -7.0 | -2.2 (7.3)
  Day 4 (72 hours post-dose) | 1.2 (3.9) | -6.0 | 1.0 (11.2)
  Day 5 (96 hours post-dose) | -0.5 (5.7) | -4.0 | -2.4 (13.8)
  Day 12 | -1.5 (6.0) | -1.0 | -1.4 (10.3)

26. Secondary Outcome: Mean Change in the Electrocardiogram (ECG) Corrected QT Interval by Fridericia (QTcF) Interval From Baseline
Description: as for outcome 13
Time Frame: Day 5
Population: The safety analysis population set included all participants who receive any amount of study product.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
Number analyzed (Participants) | 6 | 1 | 5
ms | 5.3 (13.3) | 25.0 | -10.0 (10.9)

ADVERSE EVENTS:
Time Frame: Participants were assessed for SAEs and all cause mortality from the time of study product administration through Day 85. Adverse events and clinical safety laboratory events were evaluated from the first study product administration through Day 12.
Arm/Group | Healthy Matched Controls | ESRD Not on Dialysis | Severe Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/1 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/1 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Matched Controls (N=6) | ESRD Not on Dialysis (N=1) | Severe Renal Impairment (N=5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT03896750/Prot_001.pdf
  • Statistical Analysis Plan (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT03896750/SAP_002.pdf
  • Informed Consent Form (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT03896750/ICF_000.pdf